CLINICAL TRIAL: NCT06594692
Title: Node-sparing Modified Short-Course Radiation Combined with CAPOX and Sintilimab for MSS Locally Advanced Colon Cancer : a Randomized, Prospective, Multicenter, Open-label Clinical Trial
Brief Title: Node-Sparing Short-Course Radiation with CAPOX and Sintilimab for MSS Locally Advanced Colon Cancer: a Randomized, Prospective, Multicenter Study
Acronym: mRCAT-C
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Zhangfa Song, Professor, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mRCAT-C
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Microsatellite Stable (MSS) Colon Cancer; Locally Advanced Colon Cancer
Keywords: Locally Advanced Colon Cancer; Microsatellite Stable (MSS) Colon Cancer; Node-Sparing Radiotherapy; Short-Course Radiotherapy; Sintilimab
MeSH Terms: conditions — Spinocerebellar Degenerations; Colonic Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Node-Sparing Short-Course Radiotherapy Combined with CAPOX and Sintilimab (Experimental): Intervention Procedure:
  1. Radiotherapy: Short-course radiotherapy is administered, with a total dose of 25Gy (5Gy per session for 5 sessions) targeting the primary tumor.
  2. Chemotherapy and Immunotherapy: On the 8th day after the start of radiotherapy, CAPOX chemotherapy combined with Sintilimab is initiated for 4 cycles.
  3. Surgery: One week after the completion of chemotherapy and immunotherapy, patients will undergo radical total mesorectal excision surgery.
  4. Postoperative Adjuvant Chemotherapy: Starting 3-4 weeks after surgery, patients will resume CAPOX chemotherapy for an additional 4 cycles as adjuvant treatment.
  Interventions: Drug: Node-Sparing Short-Course Radiotherapy Combined with CAPOX and Sintilimab
- Preoperative CAPOX Regimen as Neoadjuvant Therapy (Active Comparator): Intervention Procedure:
  1. Chemotherapy: Administer CAPOX chemotherapy for 4 cycles.
  2. Surgery: One week after the completion of chemotherapy, patients will undergo radical total mesorectal excision surgery.
  3. Postoperative Adjuvant Chemotherapy: Starting 3-4 weeks after surgery, patients will resume CAPOX chemotherapy for an additional 4 cycles as adjuvant treatment.
  Interventions: Drug: CAPOX Chemotherapy

INTERVENTIONS:
Drug: Node-Sparing Short-Course Radiotherapy Combined with CAPOX and Sintilimab — Radiotherapy Protocol:
  Short-course radiotherapy using three-dimensional conformal or intensity-modulated radiation therapy techniques. The radiation field will be limited to the tumor bed of the primary colon lesion, excluding surrounding draining lymph nodes and enlarged lymph nodes. The dose is fractionated as 5Gy per fraction, for a total of 25Gy over 5 fractions. Titanium clips will be placed on the proximal and distal ends of the colonic lesion via colonoscopy to guide radiation therapy positioning.
  Chemotherapy Protocol (CAPOX Regimen):
  1. Oxaliplatin: 130 mg/m², administered intravenously (ivgtt), on day 1 (d1).
  2. Capecitabine: 1000 mg/m², orally (po), twice daily (bid), from day 1 to day 14 (d1-14).
  Immunotherapy Protocol:
  During preoperative treatment, Sintilimab (immune checkpoint inhibitor) will be administered concurrently with each chemotherapy cycle.
  Arms: Node-Sparing Short-Course Radiotherapy Combined with CAPOX and Sintilimab
Drug: CAPOX Chemotherapy — Participants will receive 4 cycles of CAPOX chemotherapy followed by radical total mesorectal excision surgery, and then 4 additional cycles of postoperative CAPOX chemotherapy.
  Arms: Preoperative CAPOX Regimen as Neoadjuvant Therapy

SUMMARY:
This study aims to evaluate the use of node-sparing short-course radiotherapy combined with chemotherapy and Sintilimab, or chemotherapy alone, as neoadjuvant therapy for MSS-type locally advanced colon cancer. The goal is to explore the efficacy and safety of combining node-sparing short-course radiotherapy with chemotherapy and immunotherapy in the neoadjuvant setting for MSS-type locally advanced colon cancer, while also investigating the specific role of regional lymph nodes in tumor immunotherapy.

DETAILED DESCRIPTION:
Colorectal cancer is currently one of the most common malignant tumors in China. According to the latest data released by the National Cancer Center, it ranks second in incidence and fourth in mortality among all cancer types. Statistics indicate that approximately 50% of colon cancer patients in China are in stages II-III. Currently, adjuvant chemotherapy regimens containing oxaliplatin and 5-fluorouracil are the standard treatment for stage III and high-risk stage II colon cancer patients. However, under standard treatment protocols, the 5-year disease-free survival (DFS) rate for stage III colon cancer is less than 64%, with a recurrence rate exceeding 20%. Patients with higher T and N stages face a significantly increased risk of recurrence, severely impacting survival rates and imposing a substantial burden on both the healthcare system and society.

Neoadjuvant chemotherapy, which is administered before surgery, offers several theoretical advantages, including shrinking the primary tumor to improve surgical resection rates, reducing intraoperative tumor cell spread, and eliminating micrometastases and subclinical lesions to lower the risk of postoperative metastasis. However, data on neoadjuvant chemotherapy for locally advanced colon cancer remains limited. The FOxTROT study found that preoperative neoadjuvant chemotherapy significantly reduced the 2-year recurrence rate for locally advanced colon cancer, achieved tumor downstaging, and provided a 4% pathological complete response (pCR) rate. This study also demonstrated a strong correlation between pathological response to neoadjuvant therapy and recurrence risk, with patients achieving pCR or major pathological response (mPR) having significantly lower recurrence rates.

Recent studies have shown that combining immunotherapy with radiotherapy has a synergistic effect, even in MSS-type colorectal cancer patients. Radiotherapy can induce immunogenic cell death, releasing tumor-associated antigens and enhancing the function of dendritic cells, thereby increasing T-cell infiltration. Moreover, chemotherapy can alter the tumor microenvironment, promote angiogenesis, and improve oxygen distribution, further enhancing the efficacy of radiotherapy. One prospective phase II clinical trial involving locally advanced rectal cancer patients showed promising results, with a pCR rate of 46.2% in patients with proficient mismatch repair (pMMR), suggesting a favorable response to neoadjuvant therapy.

Lymph nodes, as secondary lymphoid organs, play a crucial role in tumor diagnosis and treatment. Recent preclinical studies have shown that tumor-draining lymph nodes (TDLNs) are essential in antigen activation and effector T-cell differentiation. On the other hand, tertiary lymphoid structures (TLS), which are organized immune cell aggregates formed in non-lymphoid tissues, have been associated with improved prognosis in cancer patients. However, the role of TDLNs in immunotherapy remains underexplored.

Based on these findings, the research team hypothesizes that tumor-draining lymph nodes play a positive role in immunotherapy response, and sparing these nodes during radiotherapy may enhance the efficacy of immunotherapy for MSS-type colorectal cancer. The team previously conducted a phase II clinical study (NCT04503694) investigating the safety and efficacy of node-sparing short-course radiotherapy combined with CAPOX chemotherapy and PD-1 inhibitors in MSS-type locally advanced rectal cancer. Results showed a 100% response rate to neoadjuvant therapy, with a pCR rate of 78.8% and a major pathological response (mPR) rate of 91%, while maintaining a high rate of organ preservation.

Given the high recurrence rates and treatment challenges associated with locally advanced colon cancer, and building on the promising results of previous studies, the research team intends to conduct the mRCAT-C study. This study aims to explore the clinical efficacy and safety of a node-sparing short-course radiotherapy combined with immunotherapy as a neoadjuvant treatment for MSS-type locally advanced colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients willing to undergo neoadjuvant treatment. 2. Age ≥ 18 years. 3. Tumor confirmed by colonoscopy and enhanced abdominal CT to be ≥ 12 cm from the anal verge.

  4. Histologically diagnosed adenocarcinoma; genetic testing indicates MSI-L or MSS, or immunohistochemistry from tumor biopsy shows pMMR (all four proteins-MSH1, MSH2, MSH6, and PMS2-are positive).

  5. Clinical staging by enhanced abdominal CT evaluates as cT3-4N0-2M0. 6. ECOG performance status score of 0-1. 7. No prior treatment with anti-tumor, immunotherapy, or abdominal radiation therapy before enrollment.

  8. Blood test results (without transfusion within 14 days and no use of granulocyte colony-stimulating factor or other hematopoietic stimulators within 7 days before the lab test):
  1. White blood cell count ≥ 3.5 × 10^9/L, absolute neutrophil count ≥ 1.5 × 10^9/L, platelet count ≥ 100 × 10^9/L, hemoglobin concentration ≥ 9 g/dL;
  2. Liver function tests (bilirubin ≤ 1.5 × ULN; AST and ALT ≤ 5 × ULN);
  3. Renal function (serum creatinine ≤ 1.5 × ULN or creatinine clearance (CCr) ≥ 50 mL/min);
  4. Coagulation (INR ≤ 1.5 × ULN, PT and APTT ≤ 1.5 × ULN);
  5. Thyroid function: TSH ≤ upper limit of normal (ULN); if abnormal, FT3 and FT4 levels must be evaluated, and if FT3 and FT4 are normal, the patient is eligible.

     9. Voluntary participation with a signed informed consent form.

     Exclusion Criteria:
* 1. History of other malignancies within the past 5 years. 2. Patients with metastases in other locations (stage IV). 3. Patients with MSI-H or dMMR. 4. Patients with conditions such as bowel obstruction, perforation, or bleeding requiring emergency surgery.

  5. Known allergy to the study drug or any of its excipients. 6. Patients with any unstable systemic diseases, including but not limited to severe infections, uncontrolled diabetes, uncontrolled hypertension, unstable angina, cerebrovascular accidents or transient ischemic attacks, myocardial infarction, congestive heart failure, or severe illnesses requiring medication (such as arrhythmias, liver, kidney, or metabolic diseases) that are life-threatening.

  7. History of active autoimmune diseases requiring systemic treatment (e.g., disease-modifying drugs, corticosteroids, or immunosuppressants) within the last 2 years. Replacement therapies (e.g., thyroid hormone, insulin, or physiological corticosteroid replacement for adrenal or pituitary insufficiency) are not considered systemic treatments.

  8. Known history of HIV infection or acquired immunodeficiency syndrome (AIDS). 9. Receipt of any investigational drug (including immunotherapy) or participation in another interventional clinical study within 30 days before screening.

  10. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study; men or women unwilling to use effective contraception during the study.

  11. Vulnerable populations, including those with mental illness, cognitive impairment, or critically ill patients.

  12. Any other conditions deemed inappropriate for participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
pathological complete response rate | 2 weeks after surgery
  The tumor specimen from node-sparing neoadjuvant chemoradiotherapy combined with immunotherapy, followed by sequential CME (complete mesocolic excision) surgery, showed no presence of cancer cells or lymph node metastasis under microscopic examination (ypT0N0M0).

SECONDARY OUTCOMES:
R0 resection rate | 2 weeks after surgery
  which is the percentage of patients who undergo a surgical procedure in which the tumor is completely removed with no cancer cells detected at the margins (edges) of the resected tissue. Achieving an R0 resection is a critical goal in cancer surgery, as it indicates that all visible and microscopic tumor cells have been removed, reducing the likelihood of recurrence.
Tumor downstaging rate | 2 weeks after surgery
  The tumor downstaging rate refers to the percentage of patients whose tumors decrease in size or extent (stage) following neoadjuvant treatment, compared to their initial stage at diagnosis. Downstaging means that the tumor has responded to treatment to the point where it moves from a more advanced stage (e.g., from stage III to stage II or I), which may improve the likelihood of successful surgical removal and lead to better prognosis.
The 3-year Event-Free Survival | 3 years post-treatment
  The 3-year Event-Free Survival (EFS) refers to the percentage of patients who remain free from certain negative events-such as cancer progression, recurrence, or death-within three years after treatment. In clinical trials, EFS is a critical measure of a treatment's long-term efficacy, indicating how long patients can live without the disease worsening or other significant events occurring during the follow-up period.
Objective Response Rate | 2 weeks after surgery
  Objective Response Rate (ORR) refers to the percentage of patients in a clinical study whose cancer shows a measurable reduction in tumor size in response to treatment.
The 3-year Local Recurrence Rate | 3 years post-treatment
  The 3-year Local Recurrence Rate (LRR) refers to the percentage of patients whose cancer returns at the original tumor site or nearby lymph nodes within three years after completing treatment. This measure is important for evaluating the long-term effectiveness of a treatment in preventing the return of cancer in the localized area where it was initially detected. A lower LRR suggests better local control of the disease.
3-year Disease-Free Survival | 3 years post-treatment
  3-year Disease-Free Survival (DFS) refers to the percentage of patients who remain free from any signs or symptoms of cancer for three years after completing treatment. It measures the length of time during which patients experience no recurrence of the disease and are considered to be in remission. DFS is commonly used to assess the effectiveness of a treatment in preventing cancer from returning within a specified time frame.
3-year Overall Survival | 3 years post-treatment
  3-year Overall Survival (OS) refers to the percentage of patients who are still alive three years after the completion of treatment, regardless of whether the cancer has recurred or progressed. It is a key indicator of the effectiveness of a treatment in prolonging life. Unlike Disease-Free Survival (DFS), OS does not take into account whether the disease has returned, focusing solely on survival.
The incidence of grade III/IV adverse events | 2 weeks after surgery
  The incidence of grade III/IV adverse events refers to the percentage of patients who experience severe or life-threatening side effects (classified as grade III or IV) during a clinical trial. Grade III adverse events are considered serious but not immediately life-threatening, often requiring medical intervention, while grade IV events are life-threatening and typically require urgent medical attention. This measure is crucial for assessing the safety and tolerability of a treatment.
EORTCQLQ-C30 | 3 years post-treatment
  The EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30) is a standardized tool used to assess the quality of life of cancer patients. It contains 30 questions that cover a wide range of physical, emotional, and social aspects of well-being, including symptoms of cancer and treatment side effects, functioning (physical, role, emotional, cognitive, and social), and overall health. The questionnaire is widely used in clinical trials to evaluate how treatments impact the patient's quality of life during and after treatment.
EORTCQLQ-CR29 | 3 years post-treatment
  The EORTC QLQ-CR29 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Colorectal Cancer Module) is a supplementary module to the QLQ-C30 designed specifically to assess quality of life in patients with colorectal cancer. It includes 29 questions that focus on colorectal cancer-specific symptoms and concerns, such as bowel function, body image, and sexual functioning, in addition to the general quality of life issues covered by the QLQ-C30. This questionnaire is used in clinical studies to evaluate the impact of colorectal cancer and its treatment on patients' quality of life.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sir Run Run Shaw Hospital, Zhejiang University, Hangzhou, China
  - Sir Run Run Shaw Hospital, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Q, Zhong W, Shen X, Hao Z, Wan M, Yang X, An R, Zhu H, Cai H, Li T, Lv Y, Dong X, Chen G, Liu A, Du J. Tertiary lymphoid structures predict survival and response to neoadjuvant therapy in locally advanced rectal cancer. NPJ Precis Oncol. 2024 Mar 2;8(1):61. doi: 10.1038/s41698-024-00533-w. PMID 38431733
- [Background] Vanhersecke L, Brunet M, Guegan JP, Rey C, Bougouin A, Cousin S, Moulec SL, Besse B, Loriot Y, Larroquette M, Soubeyran I, Toulmonde M, Roubaud G, Pernot S, Cabart M, Chomy F, Lefevre C, Bourcier K, Kind M, Giglioli I, Sautes-Fridman C, Velasco V, Courgeon F, Oflazoglu E, Savina A, Marabelle A, Soria JC, Bellera C, Sofeu C, Bessede A, Fridman WH, Loarer FL, Italiano A. Mature tertiary lymphoid structures predict immune checkpoint inhibitor efficacy in solid tumors independently of PD-L1 expression. Nat Cancer. 2021 Aug;2(8):794-802. doi: 10.1038/s43018-021-00232-6. Epub 2021 Aug 12. PMID 35118423
- [Background] Rahim MK, Okholm TLH, Jones KB, McCarthy EE, Liu CC, Yee JL, Tamaki SJ, Marquez DM, Tenvooren I, Wai K, Cheung A, Davidson BR, Johri V, Samad B, O'Gorman WE, Krummel MF, van Zante A, Combes AJ, Angelo M, Fong L, Algazi AP, Ha P, Spitzer MH. Dynamic CD8+ T cell responses to cancer immunotherapy in human regional lymph nodes are disrupted in metastatic lymph nodes. Cell. 2023 Mar 16;186(6):1127-1143.e18. doi: 10.1016/j.cell.2023.02.021. PMID 36931243
- [Background] Zhang C, Zhang L, Xu T, Xue R, Yu L, Zhu Y, Wu Y, Zhang Q, Li D, Shen S, Tan D, Bai F, Zhang H. Mapping the spreading routes of lymphatic metastases in human colorectal cancer. Nat Commun. 2020 Apr 24;11(1):1993. doi: 10.1038/s41467-020-15886-6. PMID 32332722
- [Background] Lin Z, Cai M, Zhang P, Li G, Liu T, Li X, Cai K, Nie X, Wang J, Liu J, Liu H, Zhang W, Gao J, Wu C, Wang L, Fan J, Zhang L, Wang Z, Hou Z, Ma C, Yang K, Wu G, Tao K, Zhang T. Phase II, single-arm trial of preoperative short-course radiotherapy followed by chemotherapy and camrelizumab in locally advanced rectal cancer. J Immunother Cancer. 2021 Nov;9(11):e003554. doi: 10.1136/jitc-2021-003554. PMID 34725214
- [Background] Seo I, Lee HW, Byun SJ, Park JY, Min H, Lee SH, Lee JS, Kim S, Bae SU. Neoadjuvant chemoradiation alters biomarkers of anticancer immunotherapy responses in locally advanced rectal cancer. J Immunother Cancer. 2021 Mar;9(3):e001610. doi: 10.1136/jitc-2020-001610. PMID 33692216
- [Background] Theelen WSME, Peulen HMU, Lalezari F, van der Noort V, de Vries JF, Aerts JGJV, Dumoulin DW, Bahce I, Niemeijer AN, de Langen AJ, Monkhorst K, Baas P. Effect of Pembrolizumab After Stereotactic Body Radiotherapy vs Pembrolizumab Alone on Tumor Response in Patients With Advanced Non-Small Cell Lung Cancer: Results of the PEMBRO-RT Phase 2 Randomized Clinical Trial. JAMA Oncol. 2019 Sep 1;5(9):1276-1282. doi: 10.1001/jamaoncol.2019.1478. PMID 31294749
- [Background] Diaz LA Jr, Shiu KK, Kim TW, Jensen BV, Jensen LH, Punt C, Smith D, Garcia-Carbonero R, Benavides M, Gibbs P, de la Fourchardiere C, Rivera F, Elez E, Le DT, Yoshino T, Zhong WY, Fogelman D, Marinello P, Andre T; KEYNOTE-177 Investigators. Pembrolizumab versus chemotherapy for microsatellite instability-high or mismatch repair-deficient metastatic colorectal cancer (KEYNOTE-177): final analysis of a randomised, open-label, phase 3 study. Lancet Oncol. 2022 May;23(5):659-670. doi: 10.1016/S1470-2045(22)00197-8. Epub 2022 Apr 12. PMID 35427471
- [Background] Cercek A, Lumish M, Sinopoli J, Weiss J, Shia J, Lamendola-Essel M, El Dika IH, Segal N, Shcherba M, Sugarman R, Stadler Z, Yaeger R, Smith JJ, Rousseau B, Argiles G, Patel M, Desai A, Saltz LB, Widmar M, Iyer K, Zhang J, Gianino N, Crane C, Romesser PB, Pappou EP, Paty P, Garcia-Aguilar J, Gonen M, Gollub M, Weiser MR, Schalper KA, Diaz LA Jr. PD-1 Blockade in Mismatch Repair-Deficient, Locally Advanced Rectal Cancer. N Engl J Med. 2022 Jun 23;386(25):2363-2376. doi: 10.1056/NEJMoa2201445. Epub 2022 Jun 5. PMID 35660797
- [Background] Yuan Y, Xiao WW, Xie WH, Cai PQ, Wang QX, Chang H, Chen BQ, Zhou WH, Zeng ZF, Wu XJ, Liu Q, Li LR, Zhang R, Gao YH. Neoadjuvant chemoradiotherapy for patients with unresectable radically locally advanced colon cancer: a potential improvement to overall survival and decrease to multivisceral resection. BMC Cancer. 2021 Feb 19;21(1):179. doi: 10.1186/s12885-021-07894-6. PMID 33607964
- [Background] Chang H, Yu X, Xiao WW, Wang QX, Zhou WH, Zeng ZF, Ding PR, Li LR, Gao YH. Neoadjuvant chemoradiotherapy followed by surgery in patients with unresectable locally advanced colon cancer: a prospective observational study. Onco Targets Ther. 2018 Jan 17;11:409-418. doi: 10.2147/OTT.S150367. eCollection 2018. PMID 29398921
- [Background] Qiu B, Ding PR, Cai L, Xiao WW, Zeng ZF, Chen G, Lu ZH, Li LR, Wu XJ, Mirimanoff RO, Pan ZZ, Xu RH, Gao YH. Outcomes of preoperative chemoradiotherapy followed by surgery in patients with unresectable locally advanced sigmoid colon cancer. Chin J Cancer. 2016 Jul 7;35(1):65. doi: 10.1186/s40880-016-0126-y. PMID 27389519
- [Background] Ludmir EB, Arya R, Wu Y, Palta M, Willett CG, Czito BG. Role of Adjuvant Radiotherapy in Locally Advanced Colonic Carcinoma in the Modern Chemotherapy Era. Ann Surg Oncol. 2016 Mar;23(3):856-62. doi: 10.1245/s10434-015-4907-3. Epub 2015 Oct 19. PMID 26480849
- [Background] Agas RAF, Co LBA, Sogono PG, Jacinto JCKM, Yu KKL, Jacomina LE, Bacorro WR, Sy Ortin TT. Assessing the Effect of Radiotherapy in Addition to Surgery in Colon Adenocarcinomas: a Systematic Review and Meta-analysis of Contemporary Evidence. J Gastrointest Cancer. 2020 Jun;51(2):445-460. doi: 10.1007/s12029-019-00300-2. PMID 31463890
- [Background] Fernandez LM, Sao Juliao GP, Figueiredo NL, Beets GL, van der Valk MJM, Bahadoer RR, Hilling DE, Meershoek-Klein Kranenbarg E, Roodvoets AGH, Renehan AG, van de Velde CJH, Habr-Gama A, Perez RO; International Watch & Wait Database Consortium. Conditional recurrence-free survival of clinical complete responders managed by watch and wait after neoadjuvant chemoradiotherapy for rectal cancer in the International Watch & Wait Database: a retrospective, international, multicentre registry study. Lancet Oncol. 2021 Jan;22(1):43-50. doi: 10.1016/S1470-2045(20)30557-X. Epub 2020 Dec 11. PMID 33316218
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Hu H, Zhang J, Li Y, Wang X, Wang Z, Wang H, Kang L, Liu P, Lan P, Wu X, Zhen Y, Pei H, Huang Z, Zhang H, Chen W, Zeng Y, Lai J, Wei H, Huang X, Chen J, Chen J, Tao K, Xu Q, Peng X, Liang J, Cai G, Ding K, Ding Z, Hu M, Zhang W, Tang B, Hong C, Cao J, Huang Z, Cao W, Li F, Wang X, Wang C, Huang Y, Zhao Y, Cai Y, Ling J, Xie X, Wu Z, Shi L, Ling L, Liu H, Wang J, Huang M, Deng Y; OPTICAL study group. Neoadjuvant Chemotherapy With Oxaliplatin and Fluoropyrimidine Versus Upfront Surgery for Locally Advanced Colon Cancer: The Randomized, Phase III OPTICAL Trial. J Clin Oncol. 2024 Sep 1;42(25):2978-2988. doi: 10.1200/JCO.23.01889. Epub 2024 Apr 2. PMID 38564700
- [Background] Morton D, Seymour M, Magill L, Handley K, Glasbey J, Glimelius B, Palmer A, Seligmann J, Laurberg S, Murakami K, West N, Quirke P, Gray R; FOxTROT Collaborative Group. Preoperative Chemotherapy for Operable Colon Cancer: Mature Results of an International Randomized Controlled Trial. J Clin Oncol. 2023 Mar 10;41(8):1541-1552. doi: 10.1200/JCO.22.00046. Epub 2023 Jan 19. PMID 36657089
- [Background] Hu Z, Ding J, Ma Z, Sun R, Seoane JA, Scott Shaffer J, Suarez CJ, Berghoff AS, Cremolini C, Falcone A, Loupakis F, Birner P, Preusser M, Lenz HJ, Curtis C. Quantitative evidence for early metastatic seeding in colorectal cancer. Nat Genet. 2019 Jul;51(7):1113-1122. doi: 10.1038/s41588-019-0423-x. Epub 2019 Jun 17. PMID 31209394
- [Background] van der Bij GJ, Oosterling SJ, Beelen RH, Meijer S, Coffey JC, van Egmond M. The perioperative period is an underutilized window of therapeutic opportunity in patients with colorectal cancer. Ann Surg. 2009 May;249(5):727-34. doi: 10.1097/SLA.0b013e3181a3ddbd. PMID 19387333
- [Background] Lin G, Feng Z, Liu H, Li Y, Nie Y, Liang Y, Li K. Mass screening for colorectal cancer in a population of two million older adults in Guangzhou, China. Sci Rep. 2019 Jul 18;9(1):10424. doi: 10.1038/s41598-019-46670-2. PMID 31320661
- [Background] Han B, Zheng R, Zeng H, Wang S, Sun K, Chen R, Li L, Wei W, He J. Cancer incidence and mortality in China, 2022. J Natl Cancer Cent. 2024 Feb 2;4(1):47-53. doi: 10.1016/j.jncc.2024.01.006. eCollection 2024 Mar. PMID 39036382
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204